CLINICAL TRIAL: NCT02009618
Title: The Effects of Rifaximin Therapy in Patients Pre-Diagnosed With Irritable Bowel Syndrome: A Double-Blind, Randomized, Placebo Controlled Study
Brief Title: The Effects of Rifaximin Therapy in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27.1.2013 / 1
Record Dates: First submitted 2013-11-19; First posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: IBS
Keywords: IBS; Rifaximin
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irritable bowel syndrome patients (Placebo Comparator): placebo tablet was given to another group in same doses for 10 days
  Interventions: Drug: placebo
- Rifaximin (Experimental): Irritable bowel syndrome patients
  Rifaximin is given to patients 200 mg tablets, 3x2/daily, for 10 days
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin tablet is given as 200 mg 3x2/daily, for 10 days.
  Other Names: Colidur 200 mg tablets
  Arms: Rifaximin
Drug: placebo
  Arms: Irritable bowel syndrome patients

SUMMARY:
To evaluate the efficacy of Rifaximin therapy started prior to completion of advanced examination procedure (before colonoscopy) of patients pre-diagnosed with irritable bowel syndrome, and implement it into clinical practice.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome(IBS) is a chronic relapsing disorder with unknown etiology characterized by abdominal pain and bowel habit changes without an organic pathology. Pathophysiology is not fully understood, bacterial overgrowth is one of the reasons. Because of that, use of drugs effective on the gut flora has been raised; Rifaximin is one of them. This study investigated the effectiveness of Rifaximin on IBS.

This randomized, double-blinded, controlled study began with 500 patients(144 of them removed because of incompliance). Patients those without organic bowel pathology and whom meet the Rome-III criteria, aged between 19-50 yo were enrolled in the study. Patients with known Rifaximin allergy, lactose intolerance, and those having treated for IBS whit in last 1 month as well as those with alarm symptoms (melena, fever, weight loss, anemia, rectal bleeding) were excluded. After routine biochemistry, blood count, and stool tests, Rifaximin tablet was given to a group as 1200 mg. daily in 3 divided doses, placebo tablet was given to another group in same doses for 10 days. Improvement in symptoms were scored and recorded on 10.day, 3. and 6.week. In addition to descriptive statistical methods(mean±SD), Student's-T and Mann-Whitney U-tests were used for comparison of quantitative data, chi-square and McNemar tests were used for comparison of qualitative data. Significance was accepted if p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 50 years without alarm symptoms, who were examined at the Gastroenterology Clinic, without endoscopic assessment, due to complaints of Irritable Bowel Syndrome, and pre-diagnosed with Irritable Bowel Syndrome according to the Rome III criteria, will be included in the study.

Exclusion Criteria:

1. are under the age of 18 years,
2. are allergic to Rifaximin,
3. are pregnant and lactating,
4. have documented diseases of the gastrointestinal system (such as gastric and duodenal ulcers, gastric cancer, small intestine and colon cancer, inflammatory bowel disease [Crohn's and Ulcerative Colitis], gastroparesis, chronic intestinal ischemia, etc.),
5. have (describe) documented diseases of the pancreas, biliary tract, and liver (such as pancreatitis, biliary colic pain associated with gallstones, acute cholecystitis, choledochal stone, hepatitis, hepatobiliary cancers, etc.),
6. have previously undergone major abdominal surgery,
7. have a systemic disease (such as collagen tissue disorders, kidney dysfunction, systemic infection, etc.),
8. have an identified psychiatric disorder,

   and/or
9. consume alcohol excessively

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
patients will be evaluated using a symptom severity and treatment efficacy scale after rifaximin therapy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Şentürk, Prof, Study Director — Bezmialem Vakıf University, Gastroenterology Clinic
Locations (1):
- Bezmialem Vakıf University, Gastroenterology Clinic, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Olden KW. Diagnosis of irritable bowel syndrome. Gastroenterology. 2002 May;122(6):1701-14. doi: 10.1053/gast.2002.33741. PMID 12016433
- [Background] Barbara G, De Giorgio R, Stanghellini V, Cremon C, Salvioli B, Corinaldesi R. New pathophysiological mechanisms in irritable bowel syndrome. Aliment Pharmacol Ther. 2004 Jul;20 Suppl 2:1-9. doi: 10.1111/j.1365-2036.2004.02036.x. PMID 15335408
- [Background] Talley NJ. Irritable bowel syndrome. Intern Med J. 2006 Nov;36(11):724-8. doi: 10.1111/j.1445-5994.2006.01217.x. PMID 17040359
- [Background] Majewski M, McCallum RW. Results of small intestinal bacterial overgrowth testing in irritable bowel syndrome patients: clinical profiles and effects of antibiotic trial. Adv Med Sci. 2007;52:139-42. PMID 18217406
- [Result] Schoenfeld P. Efficacy of current drug therapies in irritable bowel syndrome: what works and does not work. Gastroenterol Clin North Am. 2005 Jun;34(2):319-35, viii. doi: 10.1016/j.gtc.2005.02.002. PMID 15862938